CLINICAL TRIAL: NCT03841747
Title: A Phase II, Randomized Study of Paclitaxel Weekly Plus Pembrolizumab Versus Paclitaxel Weekly in ER-positive, Luminal B Metastatic Breast Cancer
Brief Title: Paclitaxel Plus Pembrolizumab vs. Paclitaxel Weekly in ER+ Luminal B Metastatic Breast Cancer
Acronym: PELICAN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding restrictions
Sponsor: Queen Mary University of London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012342QM; 2018-000188-10 (EudraCT Number)
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: ER-positive; Metastatic; Locally Advanced; Ki67; PAM50; Pembrolizumab; Paclitaxel; HER2-negative
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab + Paclitaxel (Experimental): 200 mg Pembrolizumab IV Q3W plus 80 mg/m2 paclitaxel IV on Days 1,8, and 15 of each 28 day cycle.
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel
- Paclitaxel (Active Comparator): 80 mg/m2 paclitaxel IV on Days 1,8, and 15 of each 28 day cycle.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg Pembrolizumab IV Q3W.
  Other Names: KEYTRUDA; lambrolizumab
  Arms: Pembrolizumab + Paclitaxel
Drug: Paclitaxel — 80 mg/m2 paclitaxel IV on Days 1,8, and 15 of each 28 day cycle.
  Other Names: Taxol

SUMMARY:
PELICAN is a randomised phase II trial that aims to evaluate the efficacy and safety of paclitaxel plus pembrolizumab relative to paclitaxel alone, in patients with locally advanced or metastatic ER-positive, HER2-negative, Luminal B breast cancer who have received no prior chemotherapy for advanced or metastatic disease.

Patients will be randomised (2:1) to one of the two treatment arms:

* Pembrolizumab plus Paclitaxel
* Paclitaxel

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Ability to comply with the protocol
3. Female ≥ 18 years of age
4. Histologically confirmed metastatic or locally advanced breast cancer that is Luminal B, ER+ve, HER2-ve.
5. Patients must have measurable disease.
6. Representative formalin-fixed paraffin embedded breast tumour samples from the primary or recurrent cancer.
7. ECOG performance status 0-1
8. Adequate haematologic and end-organ function within 28 days prior to the first study treatment
9. Patients of childbearing potential are eligible provided they have a negative serum or urine pregnancy test on Day 1 Cycle 1 (within 72 hours) of study treatment, preferably as close to the first dose as possible.

Exclusion Criteria:

1. Luminal A breast cancer
2. Prior chemotherapy for advanced or metastatic disease
3. Prior treatment with paclitaxel in the (neo)adjuvant setting within 12 months from the end of paclitaxel treatment and randomisation into this study
4. Patients with neuropathy ≥ Grade 2
5. Previous systemic treatment for other neoplasms within 5 years prior to randomisation.
6. Patients with prior allogeneic stem cell or solid organ transplantation.
7. Prior treatment with CD137 agonists, AKT inhibitors, anti-CTLA-4, anti-OX-40, anti-programmed death-1 (PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents.
8. Patients must not have a diagnosis of immunodeficiency or receiving chronic systemic steroid therapy.
9. Received therapeutic oral or intravenous antibiotics within 14 days prior to randomisation.
10. Administration of a live vaccine within 30 days prior to the first dose of study drug.
11. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL] -2) within 28days or five half-lives of the drug, whichever is shorter, prior to randomisation.
12. History of autoimmune disease.
13. History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia requiring steroids, or evidence of active pneumonitis on screening chest CT scan.
14. Active infection requiring systemic therapy.
15. History of HIV infection
16. Known active hepatitis infection.
17. Known history of active tuberculosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | At 12months
  Progression-free survival, defined as the time from the date of randomisation to the date of first documented tumour progression (using RECIST 1.1) or death from any cause, whichever occurs first.
Overall Survival | At 24 months.
  Overall Survival is defined as the time from date of randomisation to the date of death due to any cause in all patients.

SECONDARY OUTCOMES:
Objective Response Rates | Date of first documentation of CR or PR or to the date of first documented tumour progression (using RECIST 1.1) or death from any cause, whichever occurs first, assessed up to 30 months.
  Objective Response Rate is defined as the proportion of the patients in the analysis population who have a CR or PR (using RECIST 1.1).
Safety and tolerability of paclitaxel plus pembrolizumab versus paclitaxel through review of all AEs and SAEs assessed by CTCAE v4.03 | Date of randomisation to date of all adverse event resolution following discontinuation for any reason or death, assessed up to 30 months.
  Incidence, nature and severity of adverse events with severity determined according to CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, MD PhD FRCP, Principal Investigator — Queen Mary University of London